CLINICAL TRIAL: NCT05833386
Title: Effect of Preoperative Silodosin on Feasibility of Ureteral Access Sheath Insertion for Flexible Ureteroscope in Treating Renal Stones; A Prospective, Multicentre, Randomized Trial
Brief Title: Effect of Preoperative Silodosin on Feasibility of Ureteral Access Sheath Insertion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other); Alexandria University (Other); Cairo University (Other); Menoufia University (Other); Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzy Abd Elfattah Salman, Director, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pre-FURS sildosin
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silodosin group (Active Comparator): all patients will receive oral silodosin 8 mg orally for 0ne week prior to surgery
  Interventions: Procedure: Ureteral access sheath placement during flexible ureteroscope for renal stones
- Non premedicated group (Active Comparator): None of this group will receive alpha blocker prior to surgery
  Interventions: Procedure: Ureteral access sheath placement during flexible ureteroscope for renal stones

INTERVENTIONS:
Procedure: Ureteral access sheath placement during flexible ureteroscope for renal stones — Ureteral access sheath placement during flexible ureteroscope

SUMMARY:
The ureteral access sheath (UAS) is an ancillary device widely used by urologists to facilitate fast, repeatable, and safe access to ureters and collecting systems; improve visibility; reduce the risk of infection by reducing intrarenal pressure; and protect ureters and scopes when extracting multiple stones during surgery.

Insertion of ureteric access sheath may be difficult due to tight ureter, so sometimes preoperative stenting might be needed. Silodosin is an α1A adrenoceptor with high affinity and selectivity for the ureteric muscle, which may reduce ureteral spasm.

Oral a1-blockers can reduce intraureteral pressure, and may reduce maximal ureteral access sheath insertion force.¹ Preoperative silodosin protects against significant ureteral injury related to UAS insertion during fURS and decreases postoperative pain level. Silodosin premedication might be an effective and safe technique to replace prestenting.²

ELIGIBILITY:
Inclusion Criteria:

* All patients with renal stones who will undergo flexible ureteroscopy and planned for using ureteral access sheath

Exclusion Criteria:

* Paediatric age group (less than 18 year)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
failure rate of UAS insertion during FURS | 2 hours

SECONDARY OUTCOMES:
Ureteral injuries after UAS insertion | 3 hours
  Ureter wall injury will be classified according to the following five grades:
  Grade 0: No lesion or only mucosal petechiae. Grade 1: Mucosal erosion or a mucosal flap without smooth muscle injury. Grade 2: Erosion involving the mucosa and smooth muscle but sparing the adventitia.
  Grade 3: Ureteral perforation involving the full thickness of the ureteral wall, including the adventitia.
  Grade 4: Total ureteral avulsion with a complete rupture of ureteral continuity.
Post operative pain | 12 hours after surgery
  a visual analog scale (VAS) score (0 = no pain to 10 = excruciating pain) to indicate the intensity of postoperative pain 12 h after surgery.
Complications related to the procedure | 3 months
  will be graded using the modified Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Locations (1):
- Urology department - AlAzhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koo KC, Yoon JH, Park NC, Lee HS, Ahn HK, Lee KS, Kim DK, Cho KS, Chung BH, Hong CH. The Impact of Preoperative alpha-Adrenergic Antagonists on Ureteral Access Sheath Insertion Force and the Upper Limit of Force Required to Avoid Ureteral Mucosal Injury: A Randomized Controlled Study. J Urol. 2018 Jun;199(6):1622-1630. doi: 10.1016/j.juro.2017.09.173. Epub 2018 Feb 2. PMID 29410081
- [Background] Kim JK, Choi CI, Lee SH, Han JH, Shim YS, Choo MS; Young Endourological Study group. Silodosin for Prevention of Ureteral Injuries Resulting from Insertion of a Ureteral Access Sheath: A Randomized Controlled Trial. Eur Urol Focus. 2022 Mar;8(2):572-579. doi: 10.1016/j.euf.2021.03.009. Epub 2021 Mar 23. PMID 33741297
- [Background] Traxer O, Thomas A. Prospective evaluation and classification of ureteral wall injuries resulting from insertion of a ureteral access sheath during retrograde intrarenal surgery. J Urol. 2013 Feb;189(2):580-4. doi: 10.1016/j.juro.2012.08.197. Epub 2012 Oct 8. PMID 22982421